CLINICAL TRIAL: NCT00000658
Title: A Phase III Randomized Trial of Low-Dose Versus Standard-Dose mBACOD Chemotherapy With rGM-CSF for Treatment of AIDS-Associated Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 142; 11117 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: M-BACOD protocol; Granulocyte-Macrophage Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Allopurinol; Antineoplastic Agents, Combined
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Bleomycin; Vincristine; Doxorubicin; Cyclophosphamide; Allopurinol; Methotrexate; Cytarabine; Leucovorin; sargramostim; Dexamethasone

INTERVENTIONS:
Drug: Bleomycin sulfate
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride
Drug: Cyclophosphamide
Drug: Allopurinol
Drug: Methotrexate
Drug: Cytarabine
Drug: Leucovorin calcium
Drug: Sargramostim
Drug: Dexamethasone

SUMMARY:
To determine the impact of dose intensity on tumor response and survival in patients with HIV-associated non-Hodgkin's lymphoma (NHL).

HIV-infected patients are at increased risk for developing intermediate and high-grade NHL. While combination chemotherapy for aggressive B-cell NHL in the absence of immunodeficiency is highly effective, the outcome of therapy for patients with AIDS-associated NHL has been disappointing. Treatment is frequently complicated by the occurrence of multiple opportunistic infections, as well as the presence of poor bone marrow reserve, making the administration of standard doses of chemotherapy difficult. A recent study was completed using a low-dose modification of the standard mBACOD (cyclophosphamide, doxorubicin, vincristine, bleomycin, dexamethasone, methotrexate ) treatment. A 46 percent response rate was observed in patients treated with this combination of chemotherapeutic agents, with a number of durable remissions and reduced toxicity when compared to previous experience with more standard treatments. A subsequent study showed similar effectiveness using a lower dose of methotrexate administered on day 15. It is hoped that the use of sargramostim (granulocyte-macrophage colony-stimulating factor; GM-CSF) will improve bone marrow function and allow for administration of a higher dose of chemotherapy.

DETAILED DESCRIPTION:
HIV-infected patients are at increased risk for developing intermediate and high-grade NHL. While combination chemotherapy for aggressive B-cell NHL in the absence of immunodeficiency is highly effective, the outcome of therapy for patients with AIDS-associated NHL has been disappointing. Treatment is frequently complicated by the occurrence of multiple opportunistic infections, as well as the presence of poor bone marrow reserve, making the administration of standard doses of chemotherapy difficult. A recent study was completed using a low-dose modification of the standard mBACOD (cyclophosphamide, doxorubicin, vincristine, bleomycin, dexamethasone, methotrexate ) treatment. A 46 percent response rate was observed in patients treated with this combination of chemotherapeutic agents, with a number of durable remissions and reduced toxicity when compared to previous experience with more standard treatments. A subsequent study showed similar effectiveness using a lower dose of methotrexate administered on day 15. It is hoped that the use of sargramostim (granulocyte-macrophage colony-stimulating factor; GM-CSF) will improve bone marrow function and allow for administration of a higher dose of chemotherapy.

Patients are randomized to one of two treatment groups. Patients are stratified for (1) presence or absence of a prior AIDS diagnosis, (2) Karnofsky performance status of 70 or greater and lower than 70. Treatment includes prophylaxis for meningeal lymphoma and Pneumocystis carinii pneumonia. Patients on low-dose mBACOD who experience neutropenia may be given rGM-CSF until the absolute neutrophil count improves. AZT may be initiated at the completion of chemotherapy for all patients in complete remission at that time.

PER AMENDMENT 5/30/95: This trial was closed to accrual on 11/7/94 on the recommendation of the Data and Safety Monitoring Board (DSMB), because the non-significant difference in survival between the 2 treatment groups was not expected to change with further enrollment.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis with Bactrim, aerosolized pentamidine, or dapsone.

Allowed:

ddI, except when patient is also taking allopurinol.

Patients must have the following:

* Diagnosis of HIV seropositivity and non-Hodgkin's lymphoma.
* Ability to give informed consent and willingness to comply with all procedures and visit schedule.
* If between ages of 12 and 18 must receive care under direct supervision of a pediatric oncologist, and have consent of parent, guardian, or person with power of attorney.
* Participation in clinical trials of other antiretroviral agents is at the discretion of the investigator and individual patient.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active opportunistic infection, excluding Mycobacterium avium complex, requiring antibiotic therapy.
* Another prior or current malignancy, excepting curatively treated cervical or basal cell carcinoma.
* Kaposi's sarcoma if rapidly progressive, with visceral involvement, or causing peripheral edema.
* Primary central nervous system lymphoma.

Concurrent Medication:

Excluded:

* Zidovudine (AZT) or any antiretroviral agent unless allowed by investigator. ddI is allowed except when also taking allopurinol.

Systemic myelosuppressive drugs, including trimethoprim/sulfamethoxazole (T/S), pyrimethamine/sulfa, or ganciclovir.

-

Patients with the following are excluded:

* Active opportunistic infection, excluding Mycobacterium avium complex, requiring antibiotic therapy.
* Another prior or current malignancy, excepting curatively treated cervical or basal cell carcinoma.
* Kaposi's sarcoma if rapidly progressive, with visceral involvement, or causing peripheral edema.
* Primary central nervous system lymphoma.

Prior Medication:

Excluded:

* Immunomodulating agents within 2 weeks of study entry.

Prior Treatment:

Excluded:

* Chemotherapy.

Radiation therapy as outlined in protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Study Completion 1996-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L Kaplan, Study Chair; AA Levine, Study Chair; DJ Straus, Study Chair
Locations (22):
- United States (22):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Kaplan LD, Straus DJ, Testa MA, Von Roenn J, Dezube BJ, Cooley TP, Herndier B, Northfelt DW, Huang J, Tulpule A, Levine AM. Low-dose compared with standard-dose m-BACOD chemotherapy for non-Hodgkin's lymphoma associated with human immunodeficiency virus infection. National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group. N Engl J Med. 1997 Jun 5;336(23):1641-8. doi: 10.1056/NEJM199706053362304. PMID 9171066
- [Background] Kaplan L, et al. Randomized trial of standard dose mBACOD with GM-CSF vs reduced dose mBACOD for systemic HIV-associated lymphoma: ACTG 142. Proc Annu Meet Am Assoc Cancer Res. 1995;14:A818
- [Background] Straus DJ, Huang J, Testa MA, Levine AM, Kaplan LD. Prognostic factors in the treatment of human immunodeficiency virus-associated non-Hodgkin's lymphoma: analysis of AIDS Clinical Trials Group protocol 142--low-dose versus standard-dose m-BACOD plus granulocyte-macrophage colony-stimulating factor. National Institute of Allergy and Infectious Diseases. J Clin Oncol. 1998 Nov;16(11):3601-6. doi: 10.1200/JCO.1998.16.11.3601. PMID 9817281